CLINICAL TRIAL: NCT06510907
Title: Feasibility and Acceptability of Mindfulness-based Stress Reduction Program on Patients with Nocturnal Hypertension: a Pilot Randomized Controlled Trial
Brief Title: MBSR on Nocturnal Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, clinical associate professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022.593
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: hypertension; nocturnal hypertension; mindfulness; MBSR
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mindfulness-based stress reduction program on top of usual care (Experimental): Mindfulness training will be delivered through a generic 8-week MBSR.
  Interventions: Behavioral: mindfulness based stress reduction program
- Usual Care (No Intervention): Since all participants have sub-optimal daytime BP control (grade I HT), they will be given an information sheet about lifestyle treatment for HT and be advised to adhere to these lifestyle changes at recruitment by the research assistant or research nurse (to participants in both arms). For grade I HT, it is the standard clinical practice to advise non-pharmacological treatment for a few months before increasing the doses of medications. (2) There is no additional intervention provided to the standard care group. The case doctors and the patients in the standard care arm will be informed not to amend drug treatment before the ABPM at the 8-week end-point (primary end-point in future definitive RCT). In Hong Kong, patients have unlimited access to publicly-funded primary care clinics and emergency departments for any health problem. This is not limited to participants in the trial.

INTERVENTIONS:
Behavioral: mindfulness based stress reduction program — Mindfulness training will be delivered through a generic 8-week MBSR. The MBSR will consist of weekly 2-hour classes, in which the techniques to various meditations (e.g., body scan, mindful awareness of breathing, body, sounds, thoughts, emotions, and mindful movements) will be taught and discussed. Participants will be asked to meditate for ≥40 minutes every day during the 8-week program as "homework". Besides cultivating attention control and a non-judgemental stance to experience, psychoeducation about psychological stress and stress response will also be discussed during the MBSR classes. The MBSR teacher will discuss any difficulties encountered during homework meditations in every class to enhance adherence.
  Each MBSR class can have up to 25 participants. The 8-week program will be taught by a qualified MBSR teacher
  Arms: mindfulness-based stress reduction program on top of usual care

SUMMARY:
Objectives: To examine the feasibility and acceptability of treating nocturnal hypertension by mindfulness-based stress reduction program (MBSR). This will provide data essential for the main trial, which will also examine the definite effectiveness of MBSR to reduce nocturnal blood pressure (BP).

Hypothesis to be tested: MBSR and the current trial are acceptable and safe to patients with nocturnal hypertension; and future main trial is feasible in terms of recruitment, dropout rate and adherence to MBSR/BP measurements.

Design and subjects: This pilot randomized-controlled trial will recruit 76 patients with nocturnal HT (night-time Systolic BP (SBP) during sleep 120 mmHg) and stage I hypertension (awake SBP = 135-159mmHg), as detected by ambulatory blood pressure monitoring (ABPM). Participants will be allocated in 1:1 ratio by stratified block randomization (by age and presence of mood disorder) to receive MBSR (intervention group) or usual care (control group) respectively.

Instruments: ABPM/HBPM/MBSR patients' diary. Interventions: The generic 8-week MBSR will be taught by a certified MBSR teacher. Participants in MBSR arm will be asked to meditate 40 minutes every day during the interventional period.

Main outcome measures: rate of recruitment/dropout/adherence to MBSR/BP measurements Data analysis and expected results: The rate of recruitment/dropout/adherence to MBSR/BP measurements will be presented.

The acceptability of MBSR and the trial will also be assessed by patients' interviews. A high level of rate of recruitment, adherence to both MBSR and BP measurements and acceptability to MBSR are expected.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed hypertension (HT) from clinical records (with or without anti-hypertensive medications)
* nocturnal HT (night-time systolic blood pressure [SBP] during sleep ≥120 mmHg) and stage I hypertension (daytime SBP = 135-159 mmHg), as detected by 24-hour ambulatory blood pressure monitoring (ABPM)
* no change of dose and type of anti-hypertensive(s) in the prior 2 months

Exclusion Criteria:

* patients with atrial fibrillation (these patients have greater blood pressure variability)
* daytime office systolic blood pressure (BP) ≥180 mmHg or diastolic BP ≥120 mmHg (regardless of nocturnal BP)
* patients with known obstructive sleep apnoea
* history of dementia or psychotic illnesses
* patients with end-stage malignancies
* nocturnal worker, because they will have a reverse BP pattern to other participants
* patients receiving ≥3 BP medications at maximal tolerated doses
* previous participation in structured mindfulness program(s) of ≥8 weeks or regular daily meditation practices
* reported sleep time of <4 hours per day
* patients who do not agree to keep the same dose of anti-HT medications during the trial period
* patients receiving anti-coagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
rate of recruitment | over 1- year
  number of participants recruited per month during the recruitment period
feasibility of repeated ambulatory blood pressure monitoring | baseline, 8 weeks
  the proportion of patients finishing both ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
blood pressure as measured by 24-hour ambulatory blood pressure monitoring | baseline, 8 weeks
  daytime, nighttime and overall 24-hour blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- School of public health and primary care, Hong Kong, Hong Kong